CLINICAL TRIAL: NCT00291993
Title: Vasoactive Hormones During the Night in Patients With Obstructive Sleep Apnea and Healthy Controls.
Status: Completed | Type: Observational
Sponsor: Regional Hospital Holstebro (Other)
Other Study IDs: MED.RES.HOS.2004.01.PHH
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Healthy; Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Vasoactive hormones; Blood pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Obstructive sleep apnea syndrome is complicated by considerable cardiovascular morbidity and mortality, at least partly due to hypertension. Nocturnal hypoxia, hypercapnia and acidosis stimulate chemoreceptors and presumably increased secretion of vasoactive hormones which might be responsible for hypertension in these patients.

The aim of this study is to measure the secretion of vasoactive hormones at night and to analyse the relationship between vasoactive hormones, oxygen saturation and the blood pressure at night.

ELIGIBILITY:
Inclusion Criteria:

Male and female Age 20-65 Obstructive sleep apnea

Exclusion Criteria:

Drug or alcohol abuse Pregnancy or breast feeding Cancer Clinical signs or history of disease in the heart, lungs, kidney or endocrine organs Abnormal laboratory tests Albuminuria or glucosuria Aterial hypertension for healthy subjects

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Holstebro Hospital, Department of Medical Research; Pia H Hansen, MD, Principal Investigator — Holstebro Hospital, Department of Medical Research
Locations (3):
- Denmark (3):
  - Department of Medical Research, Holstebro Hospital, Holstebro, Ringkoebing County
  - Department of Medical Research, Holstebro
  - Holstebro Hospital, Department of Medical Research, Holstebro